CLINICAL TRIAL: NCT05919225
Title: Evaluation of the Impact of the MEESSI-AHF Scale on Decision Making and the Prognosis of Patients Diagnosed With Acute Heart Failure in the Emergency
Brief Title: Risk Stratification Using MEESSI-AHF Scale in ED and Impact on AHF Outcomes
Acronym: MEESSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCB/2018/0233
Record Dates: First submitted 2023-05-25; First posted 2023-06-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-05

CONDITIONS: Acute Heart Failure; Emergencies
MeSH Terms: conditions — Emergencies | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: Open-lable, multicentre, randomized, low-intervention, non-pharmacological, clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Experimental): Once AHF has been diagnosed at ED, and before decision-making about hospitalize/discharge home is taken, physicians will objectively measure the severity of decompensation, based on risk of 30-day death using MEESSI scale. As result, patient can be allocated to low, intermediate, high or very-high risk. For patients classified as low-risk, the propocol recommendation will be discharge patient to home. For patients classified as increased risk (i.e., intermediate, high or very-high risk categories), the protocol recommendation will be to hospitalize patient. Nonetheless, final decission will be left to emergency physician, and overruling (disposition against recommendation) will be allowed. For discharged patients, there is no follow up intervention planned, and it will be based on current centre protocols.For hospitalized patients, department of admission will be based on current centre protocols, with no intervention at this level.
  Interventions: Procedure: Risk stratification before decision-making about patient hospitalization or discharge
- USUAL CARE (No Intervention): Once AHF has been diagnosed at ED, emergency physicians will decide patient disposition according to their usual strategies of care, that currently do not include risk stratification. For discharged patients, there is no follow up intervention planned, and it will be based on current centre protocols. For hospitalized patients, department of admission will be based on current centre protocols, with no intervention at this level.

INTERVENTIONS:
Procedure: Risk stratification before decision-making about patient hospitalization or discharge — Once AHF has been diagnosed at ED, and before decision-making about hospitalize/discharge home is taken, physicians will objectively measure the severity of decompensation, based on risk of 30-day death using MEESSI scale. As result, patient can be allocated to low, intermediate, high or very-high risk. For patients classified as low-risk, the propocol recommendation will be discharge patient to home. For patients classified as increased risk (i.e., intermediate, high or very-high risk categories), the protocol recommendation will be to hospitalize patient. Nonetheless, final decission will be left to emergency physician, and overruling (disposition against recommendation) will be allowed.
  Arms: INTERVENTION

SUMMARY:
Evaluate the impact the application of the MESSI-AHF scale (a risk stratification scale specifically derived and validated in patients diagnosed with acute heart failure, AHF) in decision making (admission vs. discharge) by emergency physicians in emergency departments (ED) and its potential impact on on the short-term prognosis of patients with AHF.

DETAILED DESCRIPTION:
Study 1: A non-intervention study involving the consecutive inclusion of 3,200 patients with AHF in 16 Spanish EDs managed according to the usual practice. Individual risk will be retrospectively stratified according to the MEESSI-AHF scale, and we will analyze the distribution of the categories of risk in patients admitted and discharged and the prognosis of patients with low risk discharged from the ED and compare the events observed in this subgroup of patients with the recommended international standards. Study 2: This is a cuasiexperimental study in 8 EDs with consecutive inclusion of 1,600 patients with AHF managed according to the usual practice (without stratification of risk, pre-phase) and 1,600 patients managed after the implementation of the MEESSI-AHF scales for risk stratification before the final decision making in the ED (post-phase). If the patient has low risk the calculator will propose discharge; for the remaining categories of risk the calculator will propose patient admission. The final decision corresponds to the attending physician and if this decision differs from what was proposed, a reason will be given. Study 3: Open multicentre (8 EDs) randomized clinical trial (1:1) comparing the results obtained in the patients randomized to usual clinical practice (1,600 patients) with those obtained in the patients randomized to the use of the MEESSI-AHF scale for risk stratification (1,600 patients) prior to decision making. The dynamics of the decision proposed by the scale will be the same as that in Study 2. Main outcomes (Studies 1, 2, 3): Death (by any cause and cardiovascular cause) at 30 days and at 1 year; combined event (revisit to the ED or hospitalization for AHF or death) at 30 days post-discharge (global analysis of all the patients with AHF stratified by categories of risk); days alive and outside the hospital at 30 days after the index event (consultation to the ED); and proportion of patients managed without hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AHF based on Framinham criteria
* NT-proBNP >300 pg/mL
* Patient able to consent

Exclusion Criteria:

* ST-elevation acute coronary syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day all cause death | Through study completion, an avarage of 1 year
  Death for any cause since patient randomization (day 0) to day 30
Days alive and out of hospital | Through study completion, an avarage of 1 year
  Number of days with patient staying out of hospital (it can be at home, et residencial nursing house, etc., but not at hospital) from randomization (day 0) to day 30.

SECONDARY OUTCOMES:
Composite endpoint withing 30 days after discharge (ED revisit due to AHF, hospitalization due to AHF or all-cause death) | Through study completion, an avarage of 1 year
  Event will be considered if patient present ED revisit due to AHF, hospitalization due to AHF or all-cause death from the time of discharge (from ED or after hospitalization, day 0) to day 30. Accordingly, patients dying during index event (in-hospital mortality) did not account for this outcome.
ED revisit due to AHF within the 30 days after discharge | Through study completion, an avarage of 1 year
  Event will be considered if patient present ED revisit due to AHF from the time of discharge (from ED or after hospitalization, day 0) to day 30. Accordingly, patients dying during index event (in-hospital mortality) did not account for this outcome.
Hospitalization due to AHF within the 30 days after discharge | Through study completion, an avarage of 1 year
  Event will be considered if patient is hospitalized due to AHF from the time of discharge (from ED or after hospitalization, day 0) to day 30. Accordingly, patients dying during index event (in-hospital mortality) did not account for this outcome.
All-cause death within the 30 days after discharge | Through study completion, an avarage of 1 year
  Event will be considered if patient dies from the time of discharge (from ED or after hospitalization, day 0) to day 30. Accordingly, patients dying during index event (in-hospital mortality) did not account for this outcome.
Proportion of patients with AHF managed without hospitalization. | Through study completion, an avarage of 1 year
  We will calcultate the percentage of patients with AHF that are entirely managed in the ED and sent home, without hospitalization

OTHER OUTCOMES:
Analysis of causes of overruling | Through study completion, an avarage of 1 year
  Causes of overruling will be analyzed
Sensitivity analysis per protocol | Through study completion, an avarage of 1 year
  All previous analyses will be made just using patients of the intervention arm that were managed according to recommendation provided after risk stratification with MEESSI scale (i.e., disregarding patients for whom recommendation was overruled by the emergency physician)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Miro, PhD, Principal Investigator — Hospital CLinic, Barcelona, Spain
Locations (19):
- Spain (19):
  - Emergency Department, Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Emergency department, Barcelona, Catalonia
  - Emergency Department, Hospital de Getafe, Getafe, Madrid
  - Emergency Department, Hospital de Móstoles, Móstoles, Madrid
  - Emergency Department, Hospital de Gandia, Gandia, Valencia
  - Emergency Department, Hospital de Albacete, Albacete
  - Emergency Department, Hospital Dr. Balmis, Alicante
  - Emergency Department, Hospital de Sant Pau, Barcelona
  - Emergency Department, Hospital del Mar, Barcelona
  - Emergency Department, Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Emergency Department, Hospital La Mancha, Ciudad Real
  - Emergency Department, Hospital Dr. Gregorio Marañón, Madrid
  - Emergency Department, Hospital Infanta Leonor, Madrid
  - Emergency Department, Hospital de Salamanca, Salamanca
  - Emergency Department, Hospital Marques de Valdecilla, Santander
  - Emergency Department, Hospital Sant Pau i Santa Tecla, Tarragona
  - Emergency Department, Hospital Dr. Peset, Valencia
  - Emergency Department, Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miro O, Rossello X, Gil V, Martin-Sanchez FJ, Llorens P, Herrero-Puente P, Jacob J, Bueno H, Pocock SJ; ICA-SEMES Research Group. Predicting 30-Day Mortality for Patients With Acute Heart Failure in the Emergency Department: A Cohort Study. Ann Intern Med. 2017 Nov 21;167(10):698-705. doi: 10.7326/M16-2726. Epub 2017 Oct 3. PMID 28973663
- [Result] Miro O, Rossello X, Gil V, Martin-Sanchez FJ, Llorens P, Herrero P, Jacob J, Lopez-Grima ML, Gil C, Lucas Imbernon FJ, Garrido JM, Perez-Dura MJ, Lopez-Diez MP, Richard F, Bueno H, Pocock SJ. The Usefulness of the MEESSI Score for Risk Stratification of Patients With Acute Heart Failure at the Emergency Department. Rev Esp Cardiol (Engl Ed). 2019 Mar;72(3):198-207. doi: 10.1016/j.rec.2018.05.002. Epub 2018 Jun 11. English, Spanish. PMID 29903688
- [Result] Miro O, Gil V, Rossello X, Martin-Sanchez FJ, Llorens P, Jacob J, Herrero P, Herrera Mateo S, Richard F, Escoda R, Fuentes M, Martin Mojarro E, Llauger L, Bueno H, Pocock S. Patients with acute heart failure discharged from the emergency department and classified as low risk by the MEESSI score (multiple risk estimate based on the Spanish emergency department scale): prevalence of adverse events and predictability. Emergencias. 2019 Feb;31(1):5-14. English, Spanish. PMID 30656867
- [Result] Wussler D, Kozhuharov N, Sabti Z, Walter J, Strebel I, Scholl L, Miro O, Rossello X, Martin-Sanchez FJ, Pocock SJ, Nowak A, Badertscher P, Twerenbold R, Wildi K, Puelacher C, du Fay de Lavallaz J, Shrestha S, Strauch O, Flores D, Nestelberger T, Boeddinghaus J, Schumacher C, Goudev A, Pfister O, Breidthardt T, Mueller C. External Validation of the MEESSI Acute Heart Failure Risk Score: A Cohort Study. Ann Intern Med. 2019 Feb 19;170(4):248-256. doi: 10.7326/M18-1967. Epub 2019 Jan 29. PMID 30690646
- [Result] Miro O, Rossello X, Gil V, Martin-Sanchez FJ, Llorens P, Herrero-Puente P, Jacob J, Pinera P, Mojarro EM, Lucas-Imbernon FJ, Llauger L, Aguera C, Lopez-Diez MP, Valero A, Bueno H, Pocock SJ; ICA-SEMES Research Group. Analysis of How Emergency Physicians' Decisions to Hospitalize or Discharge Patients With Acute Heart Failure Match the Clinical Risk Categories of the MEESSI-AHF Scale. Ann Emerg Med. 2019 Aug;74(2):204-215. doi: 10.1016/j.annemergmed.2019.03.010. Epub 2019 May 27. PMID 31147102
- [Result] Rossello X, Bueno H, Gil V, Jacob J, Javier Martin-Sanchez F, Llorens P, Herrero Puente P, Alquezar-Arbe A, Raposeiras-Roubin S, Lopez-Diez MP, Pocock S, Miro O. MEESSI-AHF risk score performance to predict multiple post-index event and post-discharge short-term outcomes. Eur Heart J Acute Cardiovasc Care. 2021 Apr 8;10(2):142-152. doi: 10.1177/2048872620934318. PMID 33609116

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT05919225/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT05919225/ICF_001.pdf